CLINICAL TRIAL: NCT03805516
Title: Central Obesity and Cancer Prevention for Chinese American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco State University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20429001
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Obesity, Abdominal; Cancer Prevention
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1. . Daily use of a Fitbit Alta HRTM to identify behavior patterns.
  2. 12 weekly SCOPP-CW educational modules delivered via WeChat.
  3. 6 bi-weekly WeChat tailored messages based on based on the participant's tracker information, personal goals, and preferences
  Interventions: Behavioral: SCOPP-CW
- Control (Active Comparator): 1. . Daily use of a Fitbit Alta HRTM to identify behavior patterns.
  2. 12 weekly non-tailored educational modules on general health topics delivered via WeChat.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: SCOPP-CW — The proposed intervention integrates the Social Cognitive Theory, use of everyday technology (WeChat), and an adaptation of an evidence-based program that is tailored to the behavior patterns, preferences, and cultures of premenopausal Chinese American women. The intervention includes three components: (1) daily tracking of physical activities, (2) 12 weekly educational modules on healthy lifestyle, physical activity, and breast cancer prevention, and (3) 6 bi-weekly tailored messages to include tips for lifestyle modification, stress management, and healthy weight maintenance based on the user's personal characteristics and behavior patterns.
  Arms: Intervention
Behavioral: Control — This is the comparative/control group for the intervention. The control group receives daily tracking of physical activity and 12 weekly non-tailored educational information on general health topics.
  Arms: Control

SUMMARY:
This project examines the feasibility of a smartphone-based intervention to reduce obesity and breast cancer risk among Chinese American women in San Francisco. The proposed intervention is to use the mobile application and an activity tracker device to promote a healthier lifestyle and physical activity. Ultimately, the findings will advance the NIH mission of enhancing health promotion and disease prevention.

DETAILED DESCRIPTION:
Cancer is the leading cause of death in women in the United States (US). Chinese Americans are the largest ethnic group among Asian Americans. Although the incidence of breast cancer, the most common cancer in women, has decreased among other U.S racial groups over the last 15 years, Chinese American women in California have experienced a significant increase of incidence of 1.1% from 1998 to 2013. Studies have found that assimilation stress and obesity are associated with increased risk for breast cancer in Chinese American women. There are no existing interventions targeted at breast cancer prevention among premenopausal mothers with abdominal obesity. Interventions tailored to an individual's cultural, lifestyle and social support system are needed to reduce obesity and breast cancer risk. A smartphone-based intervention provides a promising platform for obesity and cancer prevention. The overall goal of this project is to test the feasibility of an obesity and breast cancer prevention intervention among Chinese American women in San Francisco. The investigators will adapt the Healthy Mothers Healthy Children: Technology-Based Intervention to Prevent Obesity to reduce obesity and breast cancer risk in premenopausal women with abdominal obesity who have dependent children in San Francisco. The proposed intervention ("Smartphone-Based Cancer and Obesity Prevention Program for Chinese Women: SCOPP-CW) includes 12 weekly educational modules and six bi-weekly tailored messages delivered via WeChat, a popular private communication app used by Chinese and Chinese Americans. The investigators propose to conduct a pilot randomized control study (RCT) to assess the short-term efficacy of SCOPP-CW on abdominal obesity, breast cancer knowledge and attitudes, weight-related behaviors (food intake and physical activity), and metabolic risk (blood pressure, lipid profile, hemoglobin A1c), which are associated with breast cancer. Thus the investigators propose the following aims: (1) Aim 1: To estimate the preliminary efficacy of the SCOPP-CW intervention on the primary outcomes (i.e. waist circumference and breast cancer knowledge and attitudes) and secondary outcomes (i.e. body mass index, self-efficacy, food intake, physical activity at baseline, 3 months, and 6 months, and metabolic risk [blood pressure, hemoglobin A1C, and lipid panel]) at baseline and 6 months.

Aim 2: To assess feasibility by understanding participants' acceptance, barriers to adherence and recommendations for intervention using focus group interviews. The investigators anticipate that this intervention will have a significant impact on breast cancer prevention. The investigators plan to use the proposed pilot study's findings to conduct a larger scale randomized trial (R01) to test the long-term efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* be female
* be at least 18 years old
* have a waist circumference great than 80 cm
* own a smartphone
* be able to read Chinese and speak Mandarin
* be premenopausal
* have a child between the age of 1 and 18 years old.

Exclusion Criteria:

* are pregnant
* gave birth less than 12 months prior to enrollment date
* have a history of breast cancer
* have an acute or life-threatening disease (e.g., renal failure).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 18 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
waist circumference | Change from baseline waist measurement at 3 months and 6 months
  waist measured in centimeters by NIH waist circumference measurement protocol
breast cancer knowledge and attitudes | Change from baseline breast cancer screening knowledge score at 3 months and 6 months
  13-item self-report questionnaire measuring knowledge, attitude, and practice of breast cancer screening

SECONDARY OUTCOMES:
body mass index | change from baseline BMI at 3 months and 6 months
  Weight and height (weight [kg]/height [m])
self-efficacy | Change from baseline self-efficacy questionnaire score at 3 months and 6 months
  28-item self-report survey measuring self-efficacy on nutrition, stress management, physical activity
food intake | Change from baseline food frequency at 3 months and 6 months
  Chinese food frequency questionnaire (FFQ) includes 118 food items
physical activity | Change from baseline daily physical activity at 3 months and 6 months
  Daily tracking 10 hours awake time with a Fitbit device
blood pressure | Change from baseline blood pressure at 3 months and 6 months
  Systolic and diastolic blood pressure measured in mmHg
Hemoglobin A1C | Change from baseline hemoglobin A1C at 6 months
  Glycated hemoglobin to measure average level of blood sugar
Lipid panel | Change from baseline lipid panel at 6 months
  A blood test that measures the level of different types of fat (lipid molecules) in the blood
C-reactive protein | Change from baseline lipid panel at 6 months
  A blood test that measure the presence of inflammation in the body

OTHER OUTCOMES:
Number of uses of the tracking app | at 6 months
  Weekly number of uses of the tracking app
Frequency of accessing the 12 educational modules | at 6 months
  Weekly number of accessing the educational modules

CONTACTS AND LOCATIONS:
Overall Officials: Fang-yu Chou, PhD, Principal Investigator — San Francisco State University; Jyu-Lin Chen, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco State University, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No